CLINICAL TRIAL: NCT06465758
Title: Prognostic Recovery Observations and Guidance for Evaluating Stroke Survivors
Acronym: PROGRESS
Status: Recruiting | Type: Observational
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Prof. Massimo Filippi, Professor in Neurology and Director of Stroke Unit, Neurology and neurorehabilitation Units, IRCCS San Raffaele
Other Study IDs: PROGRESS
Record Dates: First submitted 2024-05-13; First posted 2024-06-20 (Actual); Last update posted 2024-06-20 (Actual); Status verified 2024-06

CONDITIONS: Acute Stroke; Functional Recovery; Prognostic Factors
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Acute stroke patients: Subjects admitted in the neurology unit at San Raffaele Hospital for acute stroke meeting the inclusion criteria will be enrolled in the observational study.

SUMMARY:
This research delves into the acute prognostic factors influencing functional recovery in individuals who have experienced a stroke. The objective is to describe patterns of functional recovery after a stroke and identify new, clinically significant outcomes or metrics that can serve as predictive indicators for post-stroke functional recovery.

DETAILED DESCRIPTION:
In this prospective observational study with additional procedures, the aim is to describe different patterns of recovery according to clinical characteristics identified during the early phases post stroke. All the additional procedure are functional and clinical tests or questionnaires validated and used for standard stroke clinical practice that pose no risk to the enrolled subject. This study, based at San Raffaele Hospital's stroke unit, will enrol subjects who suffer from stroke assessed in the acute phase (T0), at three-months (T1), six-month (T2) and 1-year post-stroke (T3). No intervention that can interfere with usual clinical practice will be administered between evaluations. Assessments include neurological, neuropsychological and physical therapy questionnaires along with functional tests validated and used in stroke clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18
* Haemorrhagic or ischaemic stroke confirmed by a clinical diagnosis and by brain imaging
* NIHSS item 5-6 ≥1
* 3 to 10 days post-stroke

Exclusion Criteria:

* Transient ischaemic attack
* Premorbid Modified Rankin Scale ≥ 4
* Acute orthopaedic complications
* Inability to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects suffering from acute stroke
Sampling Method: Probability Sample
Enrollment: 360 (Estimated)
Dates: Start 2024-05-21 (Actual); Primary Completion 2028-05 (Estimated); Study Completion 2029-05 (Estimated)

PRIMARY OUTCOMES:
Action Research Arm Test (ARAT) | Within 3-10 days post stroke and at the three-month, six-month and one-year follow-up
  To evaluate upper limb functional recovery. The score ranges from 0 (indicating low functional recovery) to 57 (high functional recovery).

SECONDARY OUTCOMES:
Functional Ambulation Classification (FAC) | Assessments will occur within 3-10 days post stroke and at the three-month, six-month and one-year follow-up
  To evaluate walking ability (independence). Score ranges from 0 (non-functional ambulation) to 5 (independent ambulation).
Modified Rankin Scale (MRS) | Assessments will occur within 3-10 days post stroke and at the three-month, six-month and one-year follow-up
  To evaluate global disability. The score ranges from 0 (indicating no symptoms) to 6 (indicating deceased).
Fugl-Meyer Assessment for upper and lower limb (FMA- UL and LL) | Assessments will occur within 3-10 days post stroke and at the three-month, six-month and one-year follow-up
  To evaluate motor function in the upper and lower limbs. The motor score ranges from 0 (indicating hemiplegia) to 100 points (representing normal motor performance) with 66 points allocated for the upper extremity and 34 points for the lower extremity.
Montreal Cognitive Assessment (MOCA) | Assessments will occur within 3-10 days post stroke and at the three-month, six-month and one-year follow-up
  To evaluate cognitive functions. Scores range from 0 to 30. Higher scores indicate better cognitive functions.
Hospital Anxiety and Depression Scale (HADS) | Assessments will occur within 3-10 days post stroke and at the three-month, six-month and one-year follow-up
  To evaluate levels of anxiety and depression. Scores range from 0 (normal) to 21 (abnormal).
Barthel Index (BI) | Assessments will occur within 3-10 days post stroke and at the three-month, six-month and one-year follow-up
  To evaluate activities of daily living. The score ranges from 0 (complete dependency) to 100 (complete independency).
Motricity Index (MI) | Assessments will occur within 3-10 days post stroke and at the three-month, six-month and one-year follow-up
  To assess motor impairment. The score ranges from 0 to 100, with higher scores indicating lower motor impairment.
Ashworth Scale (AS) | Assessments will occur within 3-10 days post stroke and at the three-month, six-month and one-year follow-up
  To evaluate spasticity. The scoring system ranges from 0 to 4, with higher scores indicating increased spasticity.
Medical Research Council Scale (MRC) | Assessments will occur within 3-10 days post stroke and at the three-month, six-month and one-year follow-up
  To evaluate muscle strength. The score ranges from 0 (indicating no muscle contraction) to 5 (normal muscle power). Higher scores indicate greater strength.
ABILHAND | Assessments will occur within 3-10 days post stroke and at the three-month, six-month and one-year follow-up
  To assess manual ability. Scoring: Patients are prompted to assess their perceived difficulty in task performance. Scores range from 0 (impossible to perform) to 46 (easy to perform). Higher scores indicate better manual ability.
Trunk Control Test (TCT) | Assessments will occur within 3-10 days post stroke and at the three-month, six-month and one-year follow-up
  To assess trunk and postural control. Scoring: points are earned based on performance in mobility tasks. Score ranges from 0 to 100. Higher scores reflect better trunk and postural control.
Mini Balance Evaluation Test (Mini-BESTest) | Assessments will occur within 3-10 days post stroke and at the three-month, six-month and one-year follow-up
  To assess transitions/anticipatory postural control, reactive postural control, sensory orientation and stability in gait. Scoring: points are awarded for performing balance tasks. Higher scores indicate better performance.
Timed Up and Go Test (TUG) | Assessments will occur within 3-10 days post stroke and at the three-month, six-month and one-year follow-up
  To assess mobility and dynamic balance. Scoring: time (seconds) taken to perform a mobility task. More time corresponds to worse performance.
10 Meters Walking Test (10MWT) | Assessments will occur within 3-10 days post stroke and at the three-month, six-month and one-year follow-up
  To assess gait speed. Scoring: time (seconds) to walk 10 meters. More time corresponds to worse performance.
6 Minutes Walking Test (6MWT) | Assessments will occur within 3-10 days post stroke and at the three-month, six-month and one-year follow-up
  To assess walking endurance. Scoring: distance (meters) walked in 6 minutes. More meters indicate better performance.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS San Raffaele, Milan, Italy

IPD SHARING:
Plan to Share IPD: No